CLINICAL TRIAL: NCT05348551
Title: State of Play of Telemedicine in the Follow-up of Children With Type 1 Diabetes
Brief Title: Overview of Telemedicine in Children With Type 1 Diabetes
Acronym: TLS-DID
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A02641-40
Record Dates: First submitted 2022-03-30; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Telemedicine; Diabetes Mellitus, Type 1; Children, Only
Keywords: Diabetes mellitus type 1; Children; Telemedicine
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of the proportion of pediatric patients with type 1 diabetes with access to remote monitoring

DETAILED DESCRIPTION:
In the follow-up of type 1 diabetes in children, contact with families besides the appointements with medical et paramedic staff (paediatrician, diabetologist, nurses) is very common but not well coded, start from telehealth hubs (like myDiabby), to less unofficial contact by phone or email. This is even more so widespread since generalization of continuous glucometer (freestyle, dexcom,...), which allowed a quick data transfer to the medical staff.

Some studies had shown that telemedicine in diabetes allowed a better glycemic control and a higher implication in the desease. Indeed, in 1999 already, HbA1c significant improvement was shown when patients was regularly called by a nurse (Thompson et al.). Same finding was demonstrated in Schiaffini and al. clinical trial in 2016. This trial also shown a better adhesion to the follow up into the telemedicine group. Despite all of this studies, in France, remote monitoring isn't standardised and financed, except the national experimentation ETAPES which promotes and financially supports the deployment of remote monitoring projects around the territory.

ELIGIBILITY:
Inclusion Criteria:

* Children with type 1 diabetes

Exclusion Criteria:

* No consent

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 0 to 17 years with type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 4800 (Estimated)
Dates: Start 2022-05-20 (Estimated); Primary Completion 2022-07-20 (Estimated); Study Completion 2022-07-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of the proportion of pediatric patients with access to remote monitoring | 1 day
  Proportion of pediatric patients with access to remote monitoring

SECONDARY OUTCOMES:
Description of the different means and modalities of remote monitoring for patients | 1 day
  Proportion of patients in the different modalities of remote monitoring
Description of the different means and modalities of remote monitoring for patients | 1 day
  Proportion of patients in the different objectives of remote monitoring
Evaluation of patients' (and parents') perception of telemonitoring using a scale | 1 day
  Perceived importance of this remote monitoring score using a scale from 1 (mean no importance, I could do without) to 10 (mean it's very important, I think it's essential)

CONTACTS AND LOCATIONS:
Overall Officials: Clémentine DUPUIS, Principal Investigator — University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: No